CLINICAL TRIAL: NCT04190472
Title: Intraoperative HPV Testing Evaluation: Multicenter Prospective Cohort Study
Brief Title: Intraoperative HPV Testing Evaluation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IOP VPH IOP Protocol
Record Dates: First submitted 2019-11-29; First posted 2019-12-09 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: HSIL, High Grade Squamous Intraepithelial Lesions; Recurrence
Keywords: HSIL; Follow-up; LEEP
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The HPV test is performed using the commercially available Hybrid Capture 2 (HC2) system (Qiagen, Gaithersburg, MD, USA), which analyses the presence of high-risk HPV types (16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59 and 68). If this is positive, it is followed by the CLART-HPV2 test (Genomica, Madrid, Spain), which is a polymerase chain reaction technique that allows the detection of 35 HPV genotypes. This technique detects both high-risk HPV (16, 18, 26, 31, 33, 35, 39, 45, 51, 52, 53, 56, 58, 59, 66, 68B, 73 and 82) and low-risk HPV (6, 11, 40, 42, 43, 44, 54, 61, 62, 70, 71, 72, 81, 83, 84, 85 and 89).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IOP VPH test: Immediately after the LEEP, a cervical sample is token for the IOP-HPV test
  Interventions: Diagnostic Test: IOP HPV test

INTERVENTIONS:
Diagnostic Test: IOP HPV test — Immediately after the LEEP, a cervical sample was taken for the IOP-HPV test

SUMMARY:
High-grade intraepithelial lesion/cervical intraepithelial neoplasia grade 2-3 is a premalignant cervical lesion caused by persistent high-risk human papillomavirus infection. Human papillomavirus test is a very sensitive risk marker of cervical cancer and it has been incorporated in the follow-up after high-grade intraepithelial lesion treatment. Papillomavirus test performed intraoperatively could be a beneficial approach to anticipate treatment failure, allow for early management and consequently a reduction in costs. The aim of this study is to evaluate if the IOP-HPV test has non-inferior diagnostic utility of HSIL/CIN2-3 recurrence at 24 months as the HPV test performed 6 months after treatment.

DETAILED DESCRIPTION:
Background:

High-Grade Intraepithelial Lesion/Cervical Intraepithelial Neoplasia grade 2-3 (HSIL/CIN2-3) is a premalignant cervical lesion caused by persistent high-risk Human papillomavirus (HPV) infection [1]. It is estimated that approximately 54,000 women in Spain are annually diagnosed with HSIL/CIN2-3, which represents a significant economic burden for the national health system [2]. Electrosurgical excision procedure (LEEP) is the standard treatment of HSIL/CIN2-3 [3,4]. In Spain, current national guidelines recommend control after LEEP at 6, and 24 months [5,6,7]. The HPV test is a sensitive marker of cervical cancer risk and it has been incorporated, with cytology, in the follow-up of squamous cervical intraepithelial lesion after a LEEP [8,9,10].

We recently showed that an HPV test performed intraoperatively (IOP-HPV) has a strong association with recurrent disease as well as a good diagnostic recurrence efficiency at 12 months, similar than the test performed at 6 months. Thus, IOP-HPV test could be feasible and useful to identify treatment failure earlier than conventional strategies [11]. These results are similar to those previously observed by other authors [12].

However, one of the limitations of previous studies was the sample size of patients to achieve greater statistical power and perform a non-inferiority study.

The aim of this study is to evaluate if the IOP-HPV test has non-inferior diagnostic utility of HSIL/CIN2-3 recurrence at 24 months as the HPV test performed 6 months after LEEP.

Material and methods

This is a multicenter prospective cohort study that will include patients diagnosed with HSIL/CIN2-3. This study will be carried out at the Hospital Vall d'Hebron in Barcelona (organizing center) and other National centers from June 2020 to June 2024. All patients will undergo a HPV test 3 months prior to treatment and will be followed for a period of 24 months.

Cytology samples will be interpreted by an experienced pathologist following the Bethesda System [13]. HPV test will be performed using the commercially available Hybrid Capture 2 (HC2) system. If this is positive, it will be followed by the CLART-HPV2 test, a PCR technique that will allow the detection of 35 HPV genotypes.

Colposcopy will be performed using a colposcope Olympus 500 after preparing the cervix with 5% acetic acid and lugol solution. Colposcopy findings will be described following the criteria of the International Federation for Cervical Pathology and Colposcopy (IFCPC) [14].

Prior to LEEP, the abnormal area will be delimited by acetic acid and iodinated lugol, a colposcopy will be performed prior to the application of 1 ml of 2% mepivacaine to each quadrant of the cervix.

The entire pathological area will be removed next to the transformation zone (TZ), followed by selective coagulation of the surgical bed by diathermic coagulation ball. Immediately after the LEEP, a cervical sample will be taken for the IOP-HPV test. At the end of the procedure an ECC will be performed using a Novak curette.

The cervical specimen will be processed in a standardized way: after staining with ink the surfaces (or the margins) of the piece, a paraffin block will be obtained from which a minimum of 12 sections, of the 4 quadrants will be examined. A margin will be considered affected if the lesion reaches the margin or is within 1mm.

After surgery, the follow-up will be performed according to the National Guidelines Recommendations5,6,7. Visits will be scheduled according to the margin status of the LEEP specimen: If the margins are negative, the patient will be reviewed at 6, 12 and 24 months with cytology, HPV test and colposcopy. If they are positive, a visit will be added 4 months after the procedure where an additional cervical cytology will be taken.

Patients with abnormal cytology (LSIL+) or abnormal colposcopy will undergo a CGB. When the TZ is not completely visible or no colposcopic abnormalities are identified, an ECC with Novak curette will also be performed.

High-grade recurrence will be considered either when the CGB confirmes HSIL/CIN2-3 or when the ECC shows HSIL.The criteria to perform a second treatment will be the histological confirmation of HSIL/CIN2-3 during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HSIL/CIN2-3 by colposcopy guided biopsy (CGB) or endocervical curettage (ECC) in the 3 months prior to LEEP and/or confirmation of HSIL/CIN2-3 in the pathologic study of the surgical specimen

Exclusion Criteria:

* Patients with acquired or congenital immunosuppression
* Patients undergoing chronic immunosuppressive treatments, prior treatment with LEEP
* Patients in whom HSIL/CIN2-3 was not histologically confirmed.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed of HSIL/CIN2-3 by colposcopy guided biopsy (CGB) or endocervical curettage (ECC) in the 3 months prior to LEEP and/or confirmation of HSIL/CIN2-3 in the pathologic study of the surgical specimen
Sampling Method: Probability Sample
Enrollment: 1553 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperatory HPV testing evaluation: non- inferior study of diagnostic utility of HSIL/CIN2-3 recurrence as 6-months HPV test. | 24 months of follow-up after LEEP
  Evaluate if the IOP-HPV test has non-inferior diagnostic utility of HSIL/CIN2-3 recurrence at 24 months as the HPV test performed 6 months after LEEP.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Centeno Mediavilla, PhD, Principal Investigator — Hospital Universitari Vall Hebron; Melissa Bradbury Lobato, PhD, Principal Investigator — Hospital Vall d'Hebron; Antonio Gil Moreno, PhD, Study Chair — Hospital Vall d'Hebron; Jordi Rabasa Antonijuan, PhD, Principal Investigator — Hospital Vall d'Hebron

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinto AP, Crum CP. Natural history of cervical neoplasia: defining progression and its consequence. Clin Obstet Gynecol. 2000 Jun;43(2):352-62. doi: 10.1097/00003081-200006000-00015. No abstract available. PMID 10863633
- [Background] Castellsague X, Remy V, Puig-Tintore LM, de la Cuesta RS, Gonzalez-Rojas N, Cohet C. Epidemiology and costs of screening and management of precancerous lesions of the cervix in Spain. J Low Genit Tract Dis. 2009 Jan;13(1):38-45. doi: 10.1097/LGT.0b013e318182cd89. PMID 19098605
- [Background] Paraskevaidis E, Kalantaridou SN, Paschopoulos M, Zikopoulos K, Diakomanolis E, Dalkalitsis N, Makrydimas G, Pappa L, Malamou-Mitsi V, Agnantis NJ. Factors affecting outcome after incomplete excision of cervical intraepithelial neoplasia. Eur J Gynaecol Oncol. 2003;24(6):541-3. PMID 14658599
- [Background] Fuste P, Bellosillo B, Santamaria X, Mancebo G, Marinoso L, Alameda F, Espinet B, Sole F, Serrano S, Carreras R. HPV determination in the control after LEEP due to CIN II-III: prospective study and predictive model. Int J Gynecol Pathol. 2009 Mar;28(2):120-6. doi: 10.1097/PGP.0b013e3181891459. PMID 19188824
- [Background] Arbyn M, Paraskevaidis E, Martin-Hirsch P, Prendiville W, Dillner J. Clinical utility of HPV-DNA detection: triage of minor cervical lesions, follow-up of women treated for high-grade CIN: an update of pooled evidence. Gynecol Oncol. 2005 Dec;99(3 Suppl 1):S7-11. doi: 10.1016/j.ygyno.2005.07.033. Epub 2005 Sep 9. PMID 16154623
- [Background] Kocken M, Uijterwaal MH, de Vries AL, Berkhof J, Ket JC, Helmerhorst TJ, Meijer CJ. High-risk human papillomavirus testing versus cytology in predicting post-treatment disease in women treated for high-grade cervical disease: a systematic review and meta-analysis. Gynecol Oncol. 2012 May;125(2):500-7. doi: 10.1016/j.ygyno.2012.01.015. Epub 2012 Jan 18. PMID 22266548
- [Background] Kocken M, Helmerhorst TJ, Berkhof J, Louwers JA, Nobbenhuis MA, Bais AG, Hogewoning CJ, Zaal A, Verheijen RH, Snijders PJ, Meijer CJ. Risk of recurrent high-grade cervical intraepithelial neoplasia after successful treatment: a long-term multi-cohort study. Lancet Oncol. 2011 May;12(5):441-50. doi: 10.1016/S1470-2045(11)70078-X. PMID 21530398
- [Background] Jeong NH, Lee NW, Kim HJ, Kim T, Lee KW. High-risk human papillomavirus testing for monitoring patients treated for high-grade cervical intraepithelial neoplasia. J Obstet Gynaecol Res. 2009 Aug;35(4):706-11. doi: 10.1111/j.1447-0756.2008.00989.x. PMID 19751331
- [Background] Kang WD, Oh MJ, Kim SM, Nam JH, Park CS, Choi HS. Significance of human papillomavirus genotyping with high-grade cervical intraepithelial neoplasia treated by a loop electrosurgical excision procedure. Am J Obstet Gynecol. 2010 Jul;203(1):72.e1-6. doi: 10.1016/j.ajog.2010.01.063. Epub 2010 Apr 24. PMID 20417477
- [Background] Rabasa J, Bradbury M, Sanchez-Iglesias JL, Guerrero D, Forcada C, Alcalde A, Perez-Benavente A, Cabrera S, Ramon-Cajal S, Hernandez J, Dinares C, Garcia A, Centeno C, Gil-Moreno A. Evaluation of the intraoperative human papillomavirus test as a marker of early cure at 12 months after electrosurgical excision procedure in women with cervical high-grade squamous intraepithelial lesion: a prospective cohort study. BJOG. 2020 Jan;127(1):99-105. doi: 10.1111/1471-0528.15932. Epub 2019 Sep 25. PMID 31502397
- [Background] Torne A, Fuste P, Rodriguez-Carunchio L, Alonso I, del Pino M, Nonell R, Cardona M, Rodriguez A, Castillo P, Pahisa J, Balasch J, Ramirez J, Ordi J. Intraoperative post-conisation human papillomavirus testing for early detection of treatment failure in patients with cervical intraepithelial neoplasia: a pilot study. BJOG. 2013 Mar;120(4):392-9. doi: 10.1111/1471-0528.12072. Epub 2012 Nov 27. PMID 23189989
- [Background] Solomon D, Davey D, Kurman R, Moriarty A, O'Connor D, Prey M, Raab S, Sherman M, Wilbur D, Wright T Jr, Young N; Forum Group Members; Bethesda 2001 Workshop. The 2001 Bethesda System: terminology for reporting results of cervical cytology. JAMA. 2002 Apr 24;287(16):2114-9. doi: 10.1001/jama.287.16.2114. PMID 11966386
- [Background] Bornstein J, Bentley J, Bosze P, Girardi F, Haefner H, Menton M, Perrotta M, Prendiville W, Russell P, Sideri M, Strander B, Tatti S, Torne A, Walker P. 2011 colposcopic terminology of the International Federation for Cervical Pathology and Colposcopy. Obstet Gynecol. 2012 Jul;120(1):166-72. doi: 10.1097/AOG.0b013e318254f90c. PMID 22914406
- See also: Guía de cribado del cáncer de cuello de útero en España, 2014. Editado por Asociación Española de Patología Cervical y Colposcopia ISBN: 978-84-608-36551. — http://www.aepcc.org/wp-content/uploads/2016/01/AEPCC_revista02.pdf